CLINICAL TRIAL: NCT01373372
Title: CRH Responsiveness in Children With Functional Dyspepsia: A Pilot Study
Brief Title: Corticotropin Releasing Hormone (CRH) Responsiveness in Children With Functional Dyspepsia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not obtained.
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Craig A. Friesen, MD, Principal Investigator, Children's Mercy Hospital Kansas City
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11 05-069
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Functional Dyspepsia
Keywords: functional dyspepsia; GI
MeSH Terms: interventions — corticorelin ovine; Corticotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Functional Dyspepsia cohort (Experimental): Cohort of subjects with functional dyspepsia
  Interventions: Drug: Acthrel
- Control cohort (Other): Control group of subjects with no functional dyspepsia
  Interventions: Drug: Acthrel

INTERVENTIONS:
Drug: Acthrel — Powder for reconstitution, 1.0 mcg/kg body weight to a maximum of 100 mcg, delivered one time via IV over one minute.
  Other Names: Corticorelin

SUMMARY:
Chronic abdominal pain is the most common persistent pain condition in children and adolescents, affecting 10-15% of children at any given time. One of the most often diagnosed types of abdominal pain is functional dyspepsia (FD). FD is an abdominal pain or discomfort (e.g., nausea, bloating) in the upper abdomen that does not get better by going to the bathroom.

For some people it appears that stress can make FD worse. In adults, stress can cause the release of a hormone called corticotropin releasing hormone (CRH). The release of CRH can cause abdominal pain by affecting how fast things move through a person's stomach and intestines. This makes the organs in the abdomen more sensitive to pain, causing tenderness of the inside lining of the stomach and intestines.

Different people react differently when the body releases CRH. Some people have abdominal pain without feeling any stress or anxiety while other people who have a lot of stress or anxiety don't have any abdominal pain. Some people have neither stress, anxiety, or abdominal pain when CRH is released into the body.

In order to see how the bodies of children with functional dyspepsia and those without functional dyspepsia react to CRH, we will do a CRH stimulation test. A CRH stimulation test is routinely done in endocrine patients. It is not routinely done for patients with functional dyspepsia or for patients who do not have functional dyspepsia.

Part of the CRH stimulation test is giving a synthetic type of corticotropin, Acthrel® (brand name for Corticorelin), as injection. Acthrel® has been approved by the Food and Drug Administration (FDA) for use.

The purpose of this research study is to see if there are differences in how the bodies of children with functional dyspepsia react to CRH versus children who don't have functional dyspepsia.

Being in this study involves one clinic visit where an IV placed and a CRH stimulation test. In this test the child will be given an injection of CRH and then observed for one hour. During that hour the child will have five blood draws through the IV and will be asked questions about their anxiety and abdominal pain. This visit will take about 4 hours.

The following things will happen:

* Your child will be asked to come to the clinic between 8a.m. and 10a.m. fasting. This means your child will have had nothing to eat or drink for 8 hours before coming to the clinic.
* If your child is a female ten years of age or older, or has started having periods, a urine pregnancy test will be done before receiving the CRH infusion.
* You and your child will each be asked to complete a survey that measures your child's anxiety.
* Your child will have a biofeedback session that will measure your child's stress. In a biofeedback session, sensors are placed on your child's fingers, wrists and forehead. These sensors are connected to a computer that monitors your child's heartbeat, skin temperature and electrical pulses on your child's skin.
* Your child will have an IV inserted into a vein in his/her arm. Your child may have a cream put on their arm to help with the pain of the IV insertion. The IV will be used to inject the CRH and draw blood. If the IV stops working and blood samples can no longer be drawn from it, your child may have another IV started or blood samples may be drawn by needle stick.
* Your child will then have 30 minutes to relax.
* Your child will then have CRH infused through the IV over one minute.
* Your child will have blood drawn through the IV five times; right before the CRH stimulation test begins and 15, 30, 45 and 60 minutes after the CRH infusion. The total amount of blood drawn for the study will be about 2 ½ tablespoons.
* Your child will be asked about their abdominal pain, nausea, bloating, stress and anxiety at three separate times during the 60 minutes.
* Your child's heart rate will be measured throughout the CRH stimulation test.

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate whether there are differences in CRH (Corticotropin Releasing Hormone) responsiveness in children and adolescents with FD (Functional Dyspepsia) as compared to controls. Further, we intend to explore relationships between CRH responsiveness, inflammatory cytokines, state and trait anxiety, and self-reported symptoms.

The specific aims of the study are:

1. To determine if changes in serum cytokine profiles, heart rate variability, stress profile parameters, state and trait anxiety, and self-reported symptoms differ between patients with FD and controls following CRH infusion.
2. To determine if changes in serum ACTH (Adreno-corticotropic Hormone) or cortisol following CRH infusion differ between patients with FD and controls or as a function of the magnitude of state or trait anxiety among FD patients.

This study is a single-site pilot study.

Biochemical response to CRH stimulation will be explored for each of the cytokines, mediators and hormones detailed herein by calculating their rate of formation, maximal concentration (Cmax), time to maximal concentration (Tmax), total body exposure (AUC) and rate of recovery (as relevant). Pharmacokinetic analyses will be applied to data where there are clear ascending and descending phases on the concentration versus time profile. Concentration versus time data will be curve fit using a peeling algorithm to generate initial polyexponential parameter estimates. Final estimates of the apparent rate of recovery will be determined from an iterative, nonlinear weighted least squares regression algorithm. Assessment of goodness of fit for the pharmacokinetic model will be made using standard criteria (e.g., Akaike and Schwartz Information Criteria, objective function and the coefficients of variation for estimated parameters), the distribution of weighted residual estimates and the association between the observed and predicted concentrations. Model-independent pharmacokinetic parameters will be calculated using standard (i.e., statistical moment theory) techniques. Individual Cmax and Tmax will be estimated by inspection of the observed plasma concentration versus time data. The area under the plasma concentration versus time curve will be determined using the mixed log-linear trapezoidal rule (no extrapolation of the AUC to infinity will be performed). These analyses will be performed in Kinetica v5.0 (ThermoElectron, Philadelphia, PA). Differences between cases and controls on continuous response variables will be compared using a two-sided independent sample t-tests. Relationships among continuous response variables will be evaluated by univariate analysis of variance, linear and nonlinear regression techniques. Categorical patient factors and response variables will be compared with the Fisher's exact test on a 2 x 2 cross-tabulation. All statistical analyses will be conducted using the SSPS software package (version 15.0, SPSS Inc., Chicago, IL).

Sample Size

A sample size of 12 for each group (controls and FD patients) was chosen. Twelve patients per group provides 99% power to detect a 1.5-fold greater ACTH secretion in FD patients as compared to controls with the standard deviation assumed to be 20% based on 2 previous adult studies (both of which detected approximately a 2-fold increase). Power may be lower for secondary analysis, however, this is considered acceptable given the pilot nature of this study.

There will be two groups consisting of subjects who have been seen in the Abdominal Pain Clinic for abdominal pain of at least 8 weeks duration and fulfilling symptom-based criteria for FD and are scheduled for endoscopy and controls, who have no recent history of abdominal pain.

Both groups will undergo the same tests/procedures.

Participants will fast for a minimum of 8 hours prior to the evaluation, which will begin between 8 and 10 AM. Female participants > 10 years of age will be given a UCG as standard practice before receiving any medication or drug. The parent and child will complete the BASC-2 and the state and trait versions of the STICSA-C. A biofeedback stress profile will be performed. Next, an IV catheter will be placed and the participant will be allowed to relax for 30 minutes prior to the next part of the study. The participant then will undergo 30 minute baseline monitoring of heart rate prior to the CRH stimulation test. Following the 30 minute baseline period, a blood sample will be obtained for serum cytokines, ACTH, cortisol, and CBG. The participant will rate the severity of abdominal pain, nausea, and bloating, respectively, on 10-point scales.

For the CRH stimulation test, corticorelin (an analogue of human CRH) will be administered at a dose of 1 mcg per kg body weight (to a maximum of 100mcg) delivered over 1 minute. Blood samples will be obtained at 15 minute intervals for 60 minutes for determination of ACTH, cortisol, and CBG concentrations. The following will be obtained or recorded at 15, 30, and 60 minutes: blood samples for cytokine concentrations, ratings (on a 10-point scale) of abdominal pain, nausea, and bloating, stress profile parameters, and self-reported state anxiety (i.e. STICSA-C Your Mood at this Moment). Heart rate monitoring will be conducted for the duration of the 60 minute period.

The CRH stimulation test is a routinely used diagnostic test in Endocrine. It is not, however, routine for either of the two groups of participants in this study.

Measures

1. Heart rate variability (HRV)

   The electrocardiogram will be recorded and HRV assessed utilizing an I-330 C2 Physiograph (J & J Engineering, Poulsbo, WA) and Window USE Physiolab software. MC-5SGW electrode cables will be used to connect to 2 wrist electrodes (+ on left) and an EDR ground which will be placed on a finger.

   The HRV signal will be derived from the ECG data. Overall power spectral analysis will be applied to the HRV signal to extract the sympathovagal parameters: power in low frequency (LF) and power in high frequency (HF). LF is defined as the area under the curve in the frequency range of 0.04-0.15 Hz and HF is defined as the area under the curve in the frequency range of 0.15-0.50 Hz. The power in the LF band (0.04-0.15 Hz) represents mainly sympathetic activity and power in the HF band (0.15-0.5 Hz) of the HRV power spectrum represents purely parasympathetic or vagal activity. The LF-to-HF ratio will also be calculated as a measure of sympathovagal balance.
2. Stress Profile

   Biofeedback stress profile readings will be recorded with a single I-330 C2 Physiograph (J & J Engineering, Poulsbo, WA), utilizing Windows USE 3 Physiolab software.

   The following modalities will be monitored on all patients:
   1. Surface Electromyograph (sEMG)- readings will be measured in microvolts (mcv) using wide band placement on the frontalis; after standard skin preparation pre-gelled silver/silver chloride Red Dot patch sensors will placed a finger's width above each eyebrow, and attached to an MV-1L sEMG cable via CL 50 alligator clips. sEMG sensors also will be placed on the pulse points on both wrists to monitor and feedback heart beat.
   2. Peripheral skin temperature (TEMP)- will be measured in degrees Fahrenheit (F.) via a thermistor (RV-5 TEMP/EDR sensor) attached to the pad of the participant's middle finger (or substitute 3rd digit) on the dominant hand.
   3. Electrodermal Response (EDR)- skin conductance activity (SCA) will be measured in microohms (µohm) by an (RV-5 TEMP/EDR sensor) attached to the dominant index finger by an SE 35 EDG 8mm snap style silver/silver chloride disc imbedded in a Velcro fastener with saline based gel on the disk, to ensure skin contact.
3. Plasma Proteins (cytokines/ mediators/ hormones)

   Approximately 39 mL of blood will be collected through the IV catheter for plasma protein determinations including TNF-α, IL-4, IL-5, IL-8, eotaxin-3, MCP-1, MMP-9, ECP, MBP, cortisol, ACTH and CBG. Plasma proteins will be measured by commercially available immunoassay kits. Table 1 presents a breakdown of the amount of blood that will be collected per each time-point. Table 2 presents sample requirements and testing laboratory.
4. Free Plasma Cortisol

   Free plasma cortisol will be calculated using the following formula:

   U = √ Z2 + 0.0122 C - Z(mean)M Where U = molar concentration of unbound cortisol, C = molar concentration of total cortisol, T= molar concentration of CBG, and Z = 0.0167 + 0.182 (T-C)(mean) M

   (0.0167 and 0.182 are constants for the affinity of CBG for cortisol at 37 degrees C and the proportion of albumin-bound to unbound cortisol, respectively.)
5. BASC-2 Profile The parent and child versions of the Behavioral Assessment Scale for Children - Second Edition (BASC-2) will be completed by the participant and one parent, respectively. The BASC-2 is an objective rating system of psychological functioning in youth that provides standardized descriptions of problems and competencies. There are different versions for children (ages 8-11), adolescents (ages 12-18), and parents (different version for those with children ages 6-11 and 12 -18). (36) Raw scores are standardized as T-scores (M=50, SD=10) based on a normative sample of 3,483 children aged 4 - 18 stratified according to US Census data. Individual subscales have good reliability (internal consistency), with the exception of the Atypicality subscale on the BASC-PRS and the Somatization and Self-Reliance subscales on the BASC-SRS (r< .70). The BASC has also demonstrated criterion-related and construct validity. The T-scores for the anxiety subscales (parent- and self-report) will be used as a measure of trait anxiety for analysis.
6. STICSA-C

   The State-Trait Inventory for Cognitive and Somatic Anxiety, Child Version (STICSA-C) was adapted from the adult version of the measure, the STICSA. (37) The STICSA-C is comprised of two separate self-report scales, each with 21 items, for measuring two distinct anxiety concepts: state anxiety and trait anxiety. The latter asks children to respond to items by indicating how they feel, in general; the former asks children to respond about how they feel right now, at this very moment. Unique to the STICSA-C, items on each scale distinctly and stably assess cognitive and somatic manifestations of anxiety. Children are asked to provide their responses using a 4-point scale (i.e., from "Never" to "Almost always" on the Trait form, and from "Not at all" to Very much" on the State form). The somatic and cognitive subscales of the STICSA-C trait scale will be used as a measure of trait anxiety, while these subscales of the state scale will be used as a measure of state anxiety, in the statistical analysis.
7. GI symptom severity

   Symptom severity will be determined for pain, nausea, and bloating, respectively, on 10 point scales with 0=none and 10=most severe with the Global Response Scale.
8. Histology

For those who undergo endoscopy, routine biopsies obtained as part of usual care will be evaluated in a blinded fashion for eosinophil density. Immunohistochemistry evaluation of tissue will be performed utilizing anti-tryptase and anti-CD4. Cell densities for eosinophils, tryptase-positive cells, and CD4-positive cells, respectively, will be determined for specimens from the gastric antrum and the duodenal bulb, respectively. A minimum of five high power fields will be evaluated with the determination of mean and peak cell counts, respectively. Pathologic diagnoses will be determined by pathologist evaluation as part of routine care.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 (functional dyspepsia):
* Ages 8-17 inclusive;
* Abdominal pain of at least 8 weeks duration and fulfilling symptom-base criteria for FD;
* Scheduled for endoscopy to evaluate dyspepsia following non-response to standard acid reduction therapy;
* >20kg/45 lbs. and,
* Group 2 (Controls):
* Ages 8-17 inclusive;
* >20kg/45 lbs.

Exclusion Criteria:

* Both groups:
* Previous abdominal surgery;
* <20 kg/45 lbs.:
* Pregnancy;
* Chronic disease requiring regular medical care (e.g. diabetes mellitus, juvenile rheumatoid arthritis, cystic fibrosis, cancer); or,
* Non-English speaking.
* Controls:
* Recent history (within 6 months) of abdominal pain, nausea, vomiting, diarrhea, constipation, or bloating based on parental and self-report.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | Over 90 minutes

SECONDARY OUTCOMES:
Stress profile | over 90 minutes
  Surface Electromyograph readings, peripheral skin temperature readings, electrodermal response
plasma protein levels | change over 60 minutes
  TNF-α, IL-4, IL-5, IL-8, eotaxin-3, MCP-1, MMP-9, ECP, MBP, cortisol, ACTH and CBG levels to be obtained at time of CRH infusion and 15, 30, 45 and 60 minutes after CRH infusion
BASC 2 profile | change over 90 minutes
  To be given 30 minutes prior to CRH infusion and 15, 30 and 60 minutes after CRH infusion
STICSA-C | change over 90 minutes
  To be given 30 minutes prior to CRH infusion and 15, 30 and 60 minutes after CRH infusion.
GI symptom severity scale | change over 90 minutes
  To be given 30 minutes prior to CRH infusion and 15, 30 and 60 minutes after CRH infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Friesen, MD, Principal Investigator — Children's Mercy Hospital and Clinics
Locations (1):
- Children's Mercy Hospital and Clinics, Kansas City, Missouri, United States